CLINICAL TRIAL: NCT03664024
Title: A Phase II Trial to Investigate Genetic Markers of Response to Pembrolizumab (MK-3475, SCH 900475) Combined With Chemotherapy as a First-line Treatment for Non-Small Cell Lung Cancer (KEYNOTE-782)
Brief Title: Biomarkers of Response to Pembrolizumab Combined With Chemotherapy in Non-Small Cell Lung Cancer (KEYNOTE-782, MK-3475-782)
Acronym: KEYNOTE-782
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-782; MK-3475-782 (Other: Merck Protocol Number); 2018-002598-22 (EudraCT Number)
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Carcinoma, Non-Small-Cell Lung; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body; Adenocarcinoma | interventions — pembrolizumab; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Standard of Care (Experimental): Participants will receive standard of care pembrolizumab combined with platinum-doublet chemotherapy for 4 cycles, then pembrolizumab plus pemetrexed maintenance for up to 31 additional cycles. The platinum doublet would be pemetrexed plus the investigator's choice of either cisplatin or carboplatin.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab, 200 mg, Day 1 of each 21-day cycle (Q3W), intravenous infusion (IV), standard of care in most countries
Drug: Pemetrexed — Pemetrexed, 500 mg/m^2 infusion, standard of care, Q3W, IV
Drug: Carboplatin — Carboplatin AUC 5 mg/mL/min, IV infusion, Day 1 of each 21-day cycle for 4 cycles (Cycles 1 - 4). Investigator's choice of either cisplatin or carboplatin.
Drug: Cisplatin — Cisplatin, 75 mg/m^2, IV infusion, Day 1 of each 21-day cycle for 4 cycles (Cycles 1 - 4). Investigator's choice of either cisplatin or carboplatin.

SUMMARY:
Participants with Stage IV nonsquamous non-small cell lung cancer (NSCLC) without prior systemic treatment will be treated with standard of care pembrolizumab combined with platinum-doublet chemotherapy for 4 cycles, then pembrolizumab plus pemetrexed maintenance for up to 31 additional cycles. The platinum doublet would be pemetrexed plus the investigator's choice of either cisplatin or carboplatin. The primary objective is to evaluate if total baseline tumor mutation burden (TMB) in cell-free circulating tumor deoxyribonucleic acid (ctDNA) is predictive of objective response per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by the investigator by estimating the level of association.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically-confirmed or cytologically-confirmed diagnosis of stage IV (M1a, M1b, or M1c [AJCC 8th edition]) nonsquamous NSCLC.
* Have confirmation that epidermal growth factor receptor- (EGFR-), anaplastic lymphoma kinase- (ALK-), c-ros oncogene 1 (ROS1), or B isoform of rapidly accelerated fibrosarcoma (BRAF) directed therapy is not indicated as primary therapy. Documentation of the absence of tumor activating EGFR mutations, BRAF mutations, ALK gene rearrangements, and ROS1 gene rearrangements is required.
* Has measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Has not received prior systemic treatment for their advanced/metastatic NSCLC. Participants who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of metastatic disease.
* Have provided sufficient evaluable Stage IV, archival, solid tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion (that was not previously irradiated) for biomarker analysis (Fine Needle Aspiration [FNA] samples will not be accepted). Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 10 days prior to the first dose of study treatment.
* A male participant must agree to use contraception through the end of treatment and for at least 120 days, and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and if participant is a woman of childbearing potential (WOCBP), agrees to follow the contraceptive guidance as provided in the protocol through the end of treatment.
* Has adequate organ function.
* Has provided blood for cell-free ctDNA analysis that has been received and determined to be of sufficient quality and quantity by the designated laboratory for the primary endpoint.

Exclusion Criteria:

* Has predominantly squamous cell histology NSCLC. Mixed tumors will be categorized by the predominant cell type.
* Has small cell elements present in NSCLC tumor.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment allocation.
* Has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, peritoneal carcinomatosis.
* Has a known history of prior malignancy except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 2 years since initiation of that therapy.
* Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study intervention.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system disease.
* Has received prior therapy with a multiple programmed cell death 1 (PD-1)/ (PD-1) receptor/programmed cell death ligand 1 (PD-L1) receptor inhibitor.
* Is expected to require any other form of antineoplastic therapy while on study (including maintenance therapy with another agent for NSCLC, radiation therapy, and/or surgical resection).
* Has received a live vaccine within 30 days prior to treatment.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients or to another monoclonal antibody.
* Has a known sensitivity to any component of cisplatin, carboplatin or pemetrexed.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Is on chronic systemic steroids. Participants with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
* Is unable or unwilling to take folic acid or vitamin B12 supplementation.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with cooperating with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (15):
- United States (3):
  - University Of Colorado ( Site 0908), Aurora, Colorado
  - Harry & Jeanette Weinberg Cancer Institute ( Site 0901), Baltimore, Maryland
  - Henry Ford Health System ( Site 0903), Detroit, Michigan
- Canada (2):
  - Kingston General Hospital ( Site 0800), Kingston, Ontario
  - CISSS de la Monteregie-Centre ( Site 0801), Greenfield Park, Quebec
- Hungary (3):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet ( Site 0400), Budapest
  - Petz Aladar Megyei Oktato Korhaz ( Site 0402), Győr
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 0401), Szolnok
- Israel (2):
  - Meir Medical Center ( Site 0501), Kfar Saba
  - Chaim Sheba Medical Center ( Site 0500), Ramat Gan
- Spain (5):
  - Hospital Universitario Insular de Gran Canaria ( Site 0700), Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Puerta de Hierro ( Site 0702), Majadahonda, Madrid
  - H.U. Vall de Hebron ( Site 0701), Barcelona
  - Hospital General Universitario 12 de Octubre ( Site 0703), Madrid
  - Hospital Universitario Central de Asturias ( Site 0704), Oviedo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bar J, Esteban E, Rodriguez-Abreu D, Aix SP, Szalai Z, Felip E, Gottfried M, Provencio M, Robinson A, Fulop A, Rao SB, Camidge DR, Speranza G, Townson SM, Kobie J, Ayers M, Dettman EJ, Hunkapiller N, McDaniel R, Jung B, Burkhardt D, Mauntz R, Csoszi T. Blood tumor mutational burden and response to pembrolizumab plus chemotherapy in non-small cell lung cancer: KEYNOTE-782. Lung Cancer. 2024 Apr;190:107506. doi: 10.1016/j.lungcan.2024.107506. Epub 2024 Feb 17. PMID 38422883

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab Plus Platinum-doublet Chemotherapy: Participants received pembrolizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W) on the first day of each 21-day cycle combined with a platinum-doublet of pemetrexed 500 mg/m^2 IV infusion plus investigators choice of either carboplatin AUC 5 mg/mL/m or cisplatin 75 mg/m^2 IV Q3W for up to 4 cycles, then pembrolizumab 200 mg plus pemetrexed 500 mg/m^2 IV infusion for up to 31 additional cycles up to ~2 years.
Period: Overall Study
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy
Started | 118
Treated | 117
Completed | 0
Not Completed | 118
Not completed — Follow-up discontinued by sponsor | 34
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Death | 80

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 116
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 114
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate is the proportion of participants who have a confirmed complete response (CR) or partial response (PR). Objective response rate is assessed by investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants with missing data are considered non-responders. The percentage of participants with an ORR is presented.
Time Frame: Up to ~25 months
Population: All participants who received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy
Number analyzed (Participants) | 117
Percentage of Participants | 40.2 [31.2 to 49.6]

2. Primary Outcome: Tumor Mutation Burden (TMB) in Cell-free Circulating Tumor Deoxyribonucleic Acid (ctDNA)
Description: Cell-free ctDNA allows the exploration of tumor features from blood samples. TMB is a measure of mutational load in tumor cells and expressed as the number of somatic mutations per megabase (mut/MB) of DNA. The mean TMB in cell-free ctDNA of participants is presented.
Time Frame: Baseline (Day 1)
Population: All participants who received at least one dose of study intervention and had samples evaluable for ctDNA TMB analysis.
Measure: Mean (Standard Deviation); unit: Mut/MB
Groups:
- Pembrolizumab Plus Platinum-doublet Chemotherapy Overall: Participants received pembrolizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W) on the first day of each 21-day cycle combined with a platinum-doublet of pemetrexed 500 mg/m^2 IV infusion plus investigators choice of either carboplatin AUC 5 mg/mL/m or cisplatin 75 mg/m^2 IV Q3W for up to 4 cycles, then pembrolizumab 200 mg plus pemetrexed 500 mg/m^2 IV infusion for up to 31 additional cycles up to ~2 years. This arm includes all responders and non-responders.
- Pembrolizumab Plus Platinum-doublet Chemotherapy Responder: Participants received pembrolizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W) on the first day of each 21-day cycle combined with a platinum-doublet of pemetrexed 500 mg/m^2 IV infusion plus investigators choice of either carboplatin AUC 5 mg/mL/m or cisplatin 75 mg/m^2 IV Q3W for up to 4 cycles, then pembrolizumab 200 mg plus pemetrexed 500 mg/m^2 IV infusion for up to 31 additional cycles up to ~2 years. Participants in this arm were considered responders if they had a complete or partial response. This arm is a subset of the overall arm.
- Pembrolizumab Plus Platinum-doublet Chemotherapy Non-responder: Participants received pembrolizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W) on the first day of each 21-day cycle combined with a platinum-doublet of pemetrexed 500 mg/m^2 IV infusion plus investigators choice of either carboplatin AUC 5 mg/mL/m or cisplatin 75 mg/m^2 IV Q3W for up to 4 cycles, then pembrolizumab 200 mg plus pemetrexed 500 mg/m^2 IV infusion for up to 31 additional cycles up to ~2 years. Participants were considered non-responders if they did not have complete or partial response. This arm is a subset of the overall arm.
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy Overall | Pembrolizumab Plus Platinum-doublet Chemotherapy Responder | Pembrolizumab Plus Platinum-doublet Chemotherapy Non-responder
Number analyzed (Participants) | 101 | 42 | 59
Mut/MB | 9 (11.6) | 8 (8.3) | 10 (13.5)

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first as assessed by investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1). The Kaplan-Meier estimate of median PFS using the product-limit (Kaplan-Meier) method for censored data is presented.
Time Frame: Up to ~36 months
Population: All participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy
Number analyzed (Participants) | 117
Months | 7.2 [5.6 to 9.8]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the start of treatment to death due to any cause. The Kaplan-Meier estimate of median PFS using the product-limit (Kaplan-Meier) method for censored data is presented.
Time Frame: Up to ~36 months
Population: All participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy
Number analyzed (Participants) | 117
Months | 18.1 [13.5 to 25.6]

5. Secondary Outcome: Percentage of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experienced an AE is presented.
Time Frame: Up to ~31 months
Population: All participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy
Number analyzed (Participants) | 117
Percentage of Participants | 100

6. Secondary Outcome: Percentage of Participants Discontinuing Study Intervention Due to an AE.
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinued the study intervention due to an AE is presented.
Time Frame: Up to ~28 months
Population: All participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab Plus Platinum-doublet Chemotherapy
Number analyzed (Participants) | 117
Percentage of Participants | 38.5

ADVERSE EVENTS:
Time Frame: For All-Cause Mortality: from allocation up to ~36 months. For AEs from start of treatment up to ~31 months.
Description: All-cause mortality: All allocated participants. Adverse events: All allocated participants who received at least 1 dose of study intervention. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab + Pemetrexed + Platinum Agent: Participants received pembrolizumab 200 mg intravenous (IV) infusion every 3 weeks (Q3W) on the first day of each 21-day cycle combined with a platinum-doublet of pemetrexed 500 mg/m^2 IV infusion plus investigators choice of either carboplatin AUC 5 mg/mL/m or cisplatin 75 mg/m^2 IV Q3W for up to 4 cycles, then pembrolizumab 200 mg plus pemetrexed 500 mg/m^2 IV infusion for up to 31 additional cycles up to ~2 years.
Arm/Group | Pembrolizumab + Pemetrexed + Platinum Agent
All-Cause Mortality (participants affected / at risk) | 80/118
Serious Adverse Events (participants affected / at risk) | 60/117
Other Adverse Events (participants affected / at risk) | 114/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Pemetrexed + Platinum Agent (N=117)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Cardiotoxicity (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (3)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Device related bacteraemia (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 11 (13)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (5)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Pemetrexed + Platinum Agent (N=117)
Anaemia (Blood and lymphatic system disorders) | 72 (109)
Leukopenia (Blood and lymphatic system disorders) | 13 (16)
Neutropenia (Blood and lymphatic system disorders) | 29 (50)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (23)
Hyperthyroidism (Endocrine disorders) | 7 (8)
Hypothyroidism (Endocrine disorders) | 14 (17)
Lacrimation increased (Eye disorders) | 14 (14)
Constipation (Gastrointestinal disorders) | 21 (24)
Diarrhoea (Gastrointestinal disorders) | 27 (44)
Nausea (Gastrointestinal disorders) | 36 (44)
Vomiting (Gastrointestinal disorders) | 22 (27)
Asthenia (General disorders) | 30 (46)
Chest pain (General disorders) | 7 (9)
Fatigue (General disorders) | 25 (39)
Mucosal inflammation (General disorders) | 10 (10)
Oedema peripheral (General disorders) | 16 (19)
Pyrexia (General disorders) | 16 (25)
Pneumonia (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 13 (19)
Alanine aminotransferase increased (Investigations) | 20 (32)
Amylase increased (Investigations) | 9 (14)
Aspartate aminotransferase increased (Investigations) | 18 (33)
Blood alkaline phosphatase increased (Investigations) | 6 (7)
Blood creatinine increased (Investigations) | 17 (30)
Gamma-glutamyltransferase increased (Investigations) | 8 (10)
Neutrophil count decreased (Investigations) | 7 (8)
Weight decreased (Investigations) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 25 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 21 (25)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Dizziness (Nervous system disorders) | 10 (10)
Dysgeusia (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 9 (10)
Neuropathy peripheral (Nervous system disorders) | 7 (7)
Renal impairment (Renal and urinary disorders) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (20)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03664024/Prot_SAP_000.pdf